CLINICAL TRIAL: NCT04557709
Title: A Descriptive Study of Major Complications in Oncology Patients With Neutropenic Fever Potentially Eligible for a Hospital at Home Program
Brief Title: Major Complication Rate in Cancer Patients With Neutropenic Fever Potentially Eligible for a Hospital at Home Program
Status: Withdrawn | Type: Observational
Why Stopped: 0 participants
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-0394; NCI-2020-06606 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0394 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-09-15; First posted 2020-09-22 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (chart review): Patients' medical charts are reviewed.
  Interventions: Other: Medical Chart Review

INTERVENTIONS:
Other: Medical Chart Review — Review of medical charts
  Other Names: Chart Review

SUMMARY:
This study investigates the major complication rate in cancer patients potentially eligible for a hospital at home program for management of neutropenic fever. "Hospital at Home" is a home care program that provides acute, inpatient care in a patient's home in place of a traditional hospital stay. Learning more about the characteristics of potentially eligible patients, including reasons for inpatient admission, rates of major complications, and situations or treatments that would be difficult to deliver in an at home setting may help to inform future program development.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Estimate the major complication rate among patients potentially eligible for a hospital at home program for management of neutropenic fever.

SECONDARY OBJECTIVES:

I. Describe the demographic and clinical characteristics of patients potentially eligible for admission to a hospital at home program for management of neutropenic fever.

II. Describe situations or treatments experienced by potentially eligible patients admitted for neutropenic fever that would be difficult to accomplish in a hypothetical hospital at home program (e.g., blood transfusions, echocardiograms, computed tomography [CT] scans).

OUTLINE:

Patients' medical charts are reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to MD Anderson Cancer Center through the Emergency Center with a diagnosis of neutropenic fever between 1/1/2019 and 12/31/2019
* Be at low risk for major complications as defined by a Multinational Association for Supportive Care in Cancer (MASCC) score < 21

Exclusion Criteria:

* Reside in a nursing home
* Homelessness
* Hospice enrollment
* A secondary reason for admission to the hospital or high risk clinical feature not captured in the MASCC score that places them at high risk for major complications in a hospital at home program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to MD Anderson Cancer Center through the Emergency Center with a diagnosis of neutropenic fever between 1/1/2019 and 12/31/2019
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who experience major complications that require escalated care | 1 month
  Percentages will be presented with exact binomial 95% confidence interval. Also, will identify significant predictors of major complications (yes or no) using univariable logistic regression.

SECONDARY OUTCOMES:
Patient demographic, clinical, and psychosocial features | 1 month
  Will describe the study sample demographic, clinical, and psychosocial features. Descriptors will include frequencies, percentages, means with standard deviations, or medians with interquartile ranges, and minimum and maximum values as appropriate.
Situations or treatments experienced by potentially eligible patients admitted for neutropenic fever that would be difficult to accomplish in a hypothetical hospital at home (HaH) program | 1 month
  Will enumerate situations and treatments observed in the study sample that could not be handled optimally in the HaH environment.

CONTACTS AND LOCATIONS:
Overall Officials: Tacara N Soones, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org